CLINICAL TRIAL: NCT06045000
Title: A Phase 1 Study to Assess the Excretion Balance, Pharmacokinetics, and Metabolism of [14C]-DC-806 in Healthy Male Participants
Brief Title: Mass Balance and Pharmacokinetics (PK) of [14C]-DC-806 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DCE806102; 2023-505367-36-00 (Other: EU CT number); J5B-MC-FHAF (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: DC-806; Mass Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [14C]-DC-806 (Experimental): Participants will receive a single oral dose of unlabeled DC-806 tablets followed by DC-806 capsule containing 3.7 MBq (100 μCi) of [14C]-DC-806 on Day 1.
  Interventions: Drug: DC-806; Drug: [14C]-DC-806

INTERVENTIONS:
Drug: DC-806 — Oral tablets
Drug: [14C]-DC-806 — Oral capsules

SUMMARY:
The primary objective of this study is to investigate the rate and routes of excretion, including the mass balance, after single oral dose administration of DC-806 containing 3.7 MBq (100 μCi) of [14C]-DC-806 in urine and feces.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male.
2. Age: 18 years to 55 years, inclusive, at screening.
3. Body mass index: 18.0 kg/m^2, inclusive, at screening.
4. Weight: ≥50 kg at screening.
5. Status: healthy participants.
6. Participants must agree to use adequate contraception as described in the protocol and not donate sperm from admission to the clinical site on Day -1 until 90 days after study drug administration.
7. All prescribed medication must have been stopped at least 14 days prior to admission to the clinical site on Day -1.
8. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St John's wort) must have been stopped at least 7 days (or 5 half-lives for certain medications, whichever is longer) prior to admission to the clinical site on Day -1. Occasional use of acetaminophen/paracetamol (eg, up to 2 grams per day) is permitted during this period and throughout the study.
9. Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to screening and admission to the clinical site (including the 24-hour stay, as applicable), and during confinement at the clinical site.
10. Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, and energy drinks), and grapefruit (juice) from 48 hours (2 days) prior to admission to the clinical site on Day -1, and during confinement at the clinical site.
11. Willingness to abstain from any strenuous physical exercise from 96 hours (4 days) prior to admission on Day -1 and during confinement at the clinical site.
12. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, 12-lead electrocardiogram, and vital signs, as judged by the Investigator.
13. Willing and able to sign the Informed Consent Form.

Exclusion Criteria:

1. Employee of ICON or the Sponsor.
2. History of relevant drug and/or food allergies, in the opinion of the Investigator.
3. Irregular defecation pattern (less than once per 2 days on average), in the opinion of the Investigator.
4. Smoking more than 5 cigarettes, 1 cigar, or 1 pipe daily.
5. Unwilling or unable to abstain from tobacco products within the 48 hours (2 days) prior to screening, admission on Day -1, and during confinement in the clinical site.
6. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 1 year prior to screening.
7. Positive drug and/or alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening or admission to the clinical site on Day -1.
8. Average intake of more than 24 units of alcohol per week (clinical site standard: 1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits).
9. Positive screen for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus 1 and 2 antibodies.
10. Participation in a drug study within 30 days prior to study drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to study drug administration in the current study.
11. Donation or loss of more than 450 mL of blood within 60 days prior to study drug administration. Donation or loss of more than 1.5 liters of blood in the 10 months prior to study drug administration in the current study.
12. Significant and/or acute illness within 5 days prior to study drug administration that may impact safety assessments, in the opinion of the Investigator.
13. For a study with a radiation burden of >0.1 mSv, the participant will be excluded if he participated in another study with a radiation burden of >0.1 mSv and ≤1 mSv in the period of 1 year prior to screening; a radiation burden of >1.1 mSv and ≤2 mSv in the period of 2 years prior to screening; a radiation burden of >2.1 mSv and ≤3 mSv in the period of 3 years prior to screening, etc.
14. Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work, or during participation in a clinical study in the period of 1 year prior to screening.
15. Unsuitable veins for infusion or blood sampling as determined by the Investigator or study staff.
16. Any other condition or prior therapy that, in the Investigator's opinion, would confound or interfere with the evaluation of safety, tolerability, or PK of the study drug, interfere with study compliance, or preclude informed consent.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Renal Clearance (CLr) of DC-806 | Day 1 to Day 11
CLr of Total Radioactivity | Day 1 to Day 11
Cumulative Amount Excreted in Urine (Aeurine) of DC-806 | Day 1 to Day 11
Aeurine of Total Radioactivity | Day 1 to Day 11
Percentage of the Dose Administered Excreted in Urine (Feurine) of DC-806 | Day 1 to Day 11
Feurine of Total Radioactivity | Day 1 to Day 11
Cumulative Amount Excreted in Feces (Aefeces) of Total Radioactivity | Day 1 to Day 11
Cumulative Amount Excreted in Vomitus (Aevomitus) of Total Radioactivity | Day 1 to Day 11
Percentage of the Dose Administered Excreted in Feces (Fefeces) of Total Radioactivity | Day 1 to Day 11
Percentage of the Dose Administered Excreted in Vomitus (Fevomitus) of Total Radioactivity | Day 1 to Day 11
Total Amount Excreted in Urine, Feces, and Vomitus (Aeurine + Aefeces + Aevomitus) of Total Radioactivity | Day 1 to Day 11
Total Percentage of the Dose Administered Excreted in Urine, Feces, and Vomitus (Feurine + Fefeces + Fevomitus) of Total Radioactivity | Day 1 to Day 11
Maximum Observed Concentration (Cmax) of DC-806 in Whole Blood | Day 1 to Day 11
Cmax of DC-806 in Plasma | Day 1 to Day 11
Cmax of Total Radioactivity in Whole Blood | Day 1 to Day 11
Cmax of Total Radioactivity in Plasma | Day 1 to Day 11
Time to Cmax (tmax) of DC-806 in Whole Blood | Day 1 to Day 11
tmax of DC-806 in Plasma | Day 1 to Day 11
tmax of Total Radioactivity in Whole Blood | Day 1 to Day 11
tmax of Total Radioactivity in Plasma | Day 1 to Day 11
Area Under the Concentration-time Curve (AUC) up to Time t, where t is the Last Point with Concentrations Above the Lower Limit of Quantification (AUC0-t) of DC-806 in Whole Blood | Day 1 to Day 11
AUC0-t of DC-806 in Plasma | Day 1 to Day 11
AUC0-t of Total Radioactivity in Whole Blood | Day 1 to Day 11
AUC0-t of Total Radioactivity in Plasma | Day 1 to Day 11
AUC from time 0 to infinity (AUC0-inf) of DC-806 in Whole Blood | Day 1 to Day 11
AUC0-inf of DC-806 in Plasma | Day 1 to Day 11
AUC0-inf of Total Radioactivity in Whole Blood | Day 1 to Day 11
AUC0-inf of Total Radioactivity in Plasma | Day 1 to Day 11
Apparent Terminal Elimination Rate Constant (λz) of DC-806 in Whole Blood | Day 1 to Day 11
λz of DC-806 in Plasma | Day 1 to Day 11
λz of Total Radioactivity in Whole Blood | Day 1 to Day 11
λz of Total Radioactivity in Plasma | Day 1 to Day 11
Apparent Terminal Elimination Half-life (t1/2) of DC-806 in Whole Blood | Day 1 to Day 11
t1/2 of DC-806 in Plasma | Day 1 to Day 11
t1/2 of Total Radioactivity in Whole Blood | Day 1 to Day 11
t1/2 of Total Radioactivity in Plasma | Day 1 to Day 11
Apparent Total Clearance (CL/F) of DC-806 in Whole Blood | Day 1 to Day 11
CL/F of DC-806 in Plasma | Day 1 to Day 11
Apparent Volume of Clearance (Vz/F) of DC-806 in Whole Blood | Day 1 to Day 11
Vz/F of DC-806 in Plasma | Day 1 to Day 11
Cmax of Total Radioactivity Blood to Plasma Ratio | Day 1 to Day 11
AUC0-inf of Total Radioactivity Blood to Plasma Ratio | Day 1 to Day 11

SECONDARY OUTCOMES:
Number of Participants who Experience an Adverse Event | Up to a maximum of 25 days
Plasma, Whole Blood, Urine, and Feces Concentrations of DC-806 Major Metabolites | Day 1 to Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Phase 1 Clinic, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No